CLINICAL TRIAL: NCT06561789
Title: Efficacy of Remineralizing Potential of β-Tricalcium Phosphate Nanoparticles Versus Functionalizedβ-Tricalcium Phosphate Nanoparticles
Brief Title: Remineralization Effect of βTricalcium Phosphate Nanoparticles Versus FunctionalizedβTricalcium Phosphate Nanoparticles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aya Magdy Elsadany (Other)
Responsible Party: Sponsor-Investigator, Aya Magdy Elsadany, Assistant lecturer of oral health and prevention department at faculty of dentistry , Tanta university, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: #-P-OH-8-22-10
Record Dates: First submitted 2024-08-10; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: White Spot Lesions[Initial Caries]on Smooth Surface of Tooth

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Functionalized Nano ᵦ tricalcium phosphate particles (Experimental): The intervention is a prepared mouth wash solution for remineralization of demineralized enamel by investigator at Nano Gate institute (Egypt,cairo,elmokatm)
  Interventions: Other: Functionalized Nano ᵦ tricalcium phosphate particles
- Nano ᵦ tricalcium phosphate particles (Experimental): The intervention is a prepared mouth wash solution for remineralization of demineralized enamel by investigator at Nano Gate institute(Egypt,cairo,elmokatm)
  Interventions: Other: Nano ᵦ tricalcium phosphate particles
- sodium fluoride mouth wash (Experimental): The intervention is mouth wash solution for remineralization of demineralized enamel from Oral-B company
  Interventions: Other: sodium fluoride mouth wash
- artifacial saliva (No Intervention): it is an artificial solution that is mimic to human saliva prepared by investigator at faculty of pharmacy Tanta university

INTERVENTIONS:
Other: Functionalized Nano ᵦ tricalcium phosphate particles — The intervention is a prepared mouth wash solution for remineralization of demineralized enamel by the investigator at Nano Gate institute (Egypt,cairo,elmokatm)
  Arms: Functionalized Nano ᵦ tricalcium phosphate particles
Other: Nano ᵦ tricalcium phosphate particles — The intervention is a prepared mouth wash solution for remineralization of demineralized enamel by the investigator at Nano Gate institute (Egypt,cairo,elmokatm)
  Arms: Nano ᵦ tricalcium phosphate particles
Other: sodium fluoride mouth wash — The intervention is mouth wash solution for remineralization of demineralized enamel from Oral-B company
  Other Names: Oral-B mouth wash
  Arms: sodium fluoride mouth wash

SUMMARY:
The study collects Sixty non carious sound human permanent premolars from Tanta University's maxillofacial surgery department. The teeth are cleaned and prepared, and randomly assigned into four groups. The specimens are analyzed using an EDX analysis scanning electron microscope, and surface micro-hardness is determined using a Digital Display Vickers Micro-hardness Tester.

DETAILED DESCRIPTION:
The study involves collecting Sixty non carious sound human permanent premolars from an outpatient clinic at Tanta University's maxillofacial surgery department. The teeth are selected for their absence of caries, hypocalcification restoration, fracture fluorosis, and cracks. The teeth are cleaned and prepared for the study, including demineralization and artificial incipient enamel carious lesion preparation. The teeth are randomly assigned into four groups: functionalized Nano ᵦ tricalcium phosphate particles, Nano ᵦ tricalcium phosphate particles, sodium fluoride mouth wash, and artificial saliva. The pH of all groups is adjusted at 7. The specimens are treated in a daily pH cycling regime, with daily solution replacements. The specimens are then dried and analyzed using an Energy Dispersive X-Ray (EDX) analysis scanning electron microscope. The element content distribution of calcium and phosphorus elements is measured, and the specimens are evaluated at base line, after demineralization, and after 2, 4, and 6 weeks. Surface micro-hardness is determined using a Digital Display Vickers Micro-hardness Tester.

Data will be collected, presented, and statistically analyzed using SPSS software package system using ANOVA at a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* The selected teeth were free from caries, hypocalcification restoration, fracture fluorosis and cracks

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
concentration of calcium and phosphorous in demineralized enamel | 6 weeks
  Assessment of calcium and phosphorous using Energy Dispersive X-Ray (EDX)analysis scanning electron microscope
enamel hardness | 6 weeks
  Surface Micro-hardness will be determined using Digital Display Vickers Micro-hardness Tester* with a Vickers diamond indenter and a 20X objective lens. A load of 100g will be applied to the surface of the specimens for 20 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Aya MS Elsadany, PHD, Principal Investigator — Tanta University
Locations (1):
- Tanta university, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Background] Seyedlar RM, Rezvani M, Barari S, Imani M, Nodehi A, Atai M. Synthesis of plate-like beta-tricalcium phosphate nanoparticles and their efficiency in remineralization of incipient enamel caries. Prog Biomater. 2019 Dec;8(4):261-276. doi: 10.1007/s40204-019-00126-y. Epub 2019 Dec 7. PMID 31813116
- [Background] Karlinsey RL, Mackey AC, Walker ER, Frederick KE. Preparation, characterization and in vitro efficacy of an acid-modified beta-TCP material for dental hard-tissue remineralization. Acta Biomater. 2010 Mar;6(3):969-78. doi: 10.1016/j.actbio.2009.08.034. Epub 2009 Aug 27. PMID 19716443
- [Background] Salinovic I, Schauperl Z, Marcius M, Miletic I. The Effects of Three Remineralizing Agents on the Microhardness and Chemical Composition of Demineralized Enamel. Materials (Basel). 2021 Oct 13;14(20):6051. doi: 10.3390/ma14206051. PMID 34683643
- [Background] Sindhura V, Uloopi KS, Vinay C, Chandrasekhar R. Evaluation of enamel remineralizing potential of self-assembling peptide P11-4 on artificially induced enamel lesions in vitro. J Indian Soc Pedod Prev Dent. 2018 Oct-Dec;36(4):352-356. doi: 10.4103/JISPPD.JISPPD_255_18. PMID 30324924
- [Background] Rirattanapong P, Vongsavan K, Suratit R, Tanaiutchawoot N, Charoenchokdilok V, Jeansuwannagorn S, Yoddee M. Effect of various forms of calcium in dental products on human enamel microhardness in vitro. Southeast Asian J Trop Med Public Health. 2012 Jul;43(4):1053-8. PMID 23077830